CLINICAL TRIAL: NCT05550805
Title: Prognostic Study of Major Adverse Cardiovascular Events in Patients With Coronary Artery Disease Based on Metabolomics, and Lipidomics
Brief Title: Prognostic Study of Major Adverse Cardiovascular Events in Patients With Coronary Artery Disease Based on Metabolomics, and Lipidomics (BIPass II)
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 20220914-Qilu
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Major Adverse Cardiovascular Events in Patients With Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate whether there were differences in metabolomics and lipidomics in patients with coronary artery disease who had major adverse cardiovascular events during follow-up compared with those who did not.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients with the diagnosis of any type of coronary artery disease;
2. Age ≥18 years of age;
3. Patient or guardian provided informed written consent.

Exclusion Criteria:

1. Prior surgery, trauma or clinically evident coagulopathic bleeding within the previous 2 weeks;
2. Bipass population with missing follow-up records in Qilu Hospital emergency follow-up cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease
Sampling Method: Probability Sample
Enrollment: 5822 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 20191101-20220701
  cardiac death, myocardial infarction, heart failure, stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Yuguo Chen, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No